CLINICAL TRIAL: NCT03234751
Title: Effect of Nesiritide Infusion on Insulin Sensitivity in Healthy Obese Insulin Resistant Subjects
Acronym: BNP3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: TRIMDFH 1081082
Record Dates: First submitted 2017-07-18; First posted 2017-07-31 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Diabetes
Keywords: human B-type natriuretic peptide
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This study is prospective randomized, double masked, 2-period cross over design, proof of concept study of the effects of intravenously administered rhBNP (nesiritide) on insulin sensitivity in otherwise healthy obese nondiabetic insulin resistant subjects.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obese nondiabetic insulin resistant subjects- Panel A (Active Comparator): IV nesiritide 3 pmol/kg/min or placebo for nesiritide
  Interventions: Drug: Continous IV infusion of Nesiritide; Drug: Hyperinsulinemic euglycemic clamp; Drug: Placebo
- Obese nondiabetic insulin resistant subjects- Panel B (Active Comparator): IV nesiritide 2 pmol/kg/min or placebo for nesiritide
  Interventions: Drug: Continous IV infusion of Nesiritide; Drug: Hyperinsulinemic euglycemic clamp; Drug: Placebo

INTERVENTIONS:
Drug: Continous IV infusion of Nesiritide — Nesiritide (fhBNP) administered by continuous IV infusion during 48 hours.
Drug: Hyperinsulinemic euglycemic clamp — 48 hours IV infusion of nesiritide on insulin sensitivity (IS) measured by two-step hyperinsulinemic euglycemic clamp in obese nondiabetic insulin resistant subjects.
Drug: Placebo — 48 hours of placebo.

SUMMARY:
The purpose of the study is to compare the effects of nesiritide to placebo administered by a continuous IV infusion over 48 hours for the treatment of insulin resistance in healthy, obese, insulin resistant individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-65 years inclusive
2. Men and women
3. Able to provide written, informed consent
4. Weight stable (± 3 kg) during the 3 months prior to enrollment
5. BMI ≥ 30 kg/m2; body weight ≤ 106 kg
6. Resting blood pressure ≥ 110/60 mmHg and ≤ 150/100 mmHg

Exclusion Criteria:

1. Known coronary artery disease, angina or heart failure
2. Type 1 or Type 2 Diabetes (A1c ≥ 6.5% and/or fasting plasma glucose >125mg/dL)
3. Bleeding disorders
4. Hemoglobin level < 12.5 g/dL for women; < 13.0 g/dL for men
5. Acute or chronic infections
6. Hepatitis and/or cirrhosis (AST or Alanine Aminotransferase 2.5 times upper limit of normal)
7. Severe asthma or chronic obstructive pulmonary disease
8. Renal insufficiency (creatinine > 1.6 mg/dL)
9. Prior bariatric surgery
10. Inflammatory bowel disease or malabsorption
11. Cancer within the last 3 years (except non-melanoma skin cancer or treated cervical carcinoma in situ)
12. Psychiatric or eating disorders
13. Untreated or inadequately controlled thyroid (abnormal TSH) or other endocrine disorders
14. Active rheumatoid arthritis or other inflammatory rheumatic disorder
15. Pregnant or nursing women
16. Presence of clinically significant abnormalities on electrocardiogram
17. Smoking (within the last 3 months)
18. Known hypersensitivity to nesiritide or any of its excipients
19. Poor intravenous access
20. Use of medications: a) nitrates, b) beta-blockers, c) digoxin, d) anti-diabetic agents, e) oral, injected or chronic topical steroids (inhaled steroids for mild asthma are acceptable), f) chronic use of aspirin or other non-steroidal anti-inflammatory drugs, including cyclooxygenase-2 inhibitors, g) other drugs known to affect immune or metabolic function and h) orlistat, phenteramine or other weight loss or anorectic agents.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
IV infusion of nesiritide at a 3pmol/kg rate | 48 hours
  Average changes in glucose disposal rates (GDR) and endogenous glucose production (EGP) from baseline corrected for body weight at steady state of the clamp during the high- and low-dose portions.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pratley, MD, Principal Investigator — Translational Reseach institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). State-specific prevalence of obesity among adults--United States, 2007. MMWR Morb Mortal Wkly Rep. 2008 Jul 18;57(28):765-8. PMID 18636063
- [Background] Poirier P, Giles TD, Bray GA, Hong Y, Stern JS, Pi-Sunyer FX, Eckel RH; American Heart Association; Obesity Committee of the Council on Nutrition, Physical Activity, and Metabolism. Obesity and cardiovascular disease: pathophysiology, evaluation, and effect of weight loss: an update of the 1997 American Heart Association Scientific Statement on Obesity and Heart Disease from the Obesity Committee of the Council on Nutrition, Physical Activity, and Metabolism. Circulation. 2006 Feb 14;113(6):898-918. doi: 10.1161/CIRCULATIONAHA.106.171016. Epub 2005 Dec 27. PMID 16380542
- [Background] Stein CJ, Colditz GA. The epidemic of obesity. J Clin Endocrinol Metab. 2004 Jun;89(6):2522-5. doi: 10.1210/jc.2004-0288. PMID 15181019
- [Background] Aneja A, El-Atat F, McFarlane SI, Sowers JR. Hypertension and obesity. Recent Prog Horm Res. 2004;59:169-205. doi: 10.1210/rp.59.1.169. PMID 14749502
- [Background] Mancia G, Bousquet P, Elghozi JL, Esler M, Grassi G, Julius S, Reid J, Van Zwieten PA. The sympathetic nervous system and the metabolic syndrome. J Hypertens. 2007 May;25(5):909-20. doi: 10.1097/HJH.0b013e328048d004. PMID 17414649
- [Background] Goodfriend TL, Kelley DE, Goodpaster BH, Winters SJ. Visceral obesity and insulin resistance are associated with plasma aldosterone levels in women. Obes Res. 1999 Jul;7(4):355-62. doi: 10.1002/j.1550-8528.1999.tb00418.x. PMID 10440591
- [Background] Sarzani R, Dessi-Fulgheri P, Paci VM, Espinosa E, Rappelli A. Expression of natriuretic peptide receptors in human adipose and other tissues. J Endocrinol Invest. 1996 Oct;19(9):581-5. doi: 10.1007/BF03349021. PMID 8957740
- [Background] Wang TJ, Larson MG, Levy D, Benjamin EJ, Leip EP, Wilson PW, Vasan RS. Impact of obesity on plasma natriuretic peptide levels. Circulation. 2004 Feb 10;109(5):594-600. doi: 10.1161/01.CIR.0000112582.16683.EA. PMID 14769680
- [Background] Potter LR, Abbey-Hosch S, Dickey DM. Natriuretic peptides, their receptors, and cyclic guanosine monophosphate-dependent signaling functions. Endocr Rev. 2006 Feb;27(1):47-72. doi: 10.1210/er.2005-0014. Epub 2005 Nov 16. PMID 16291870
- [Background] Khan AM, Cheng S, Magnusson M, Larson MG, Newton-Cheh C, McCabe EL, Coviello AD, Florez JC, Fox CS, Levy D, Robins SJ, Arora P, Bhasin S, Lam CS, Vasan RS, Melander O, Wang TJ. Cardiac natriuretic peptides, obesity, and insulin resistance: evidence from two community-based studies. J Clin Endocrinol Metab. 2011 Oct;96(10):3242-9. doi: 10.1210/jc.2011-1182. Epub 2011 Aug 17. PMID 21849523
- [Background] Chen-Tournoux A, Khan AM, Baggish AL, Castro VM, Semigran MJ, McCabe EL, Moukarbel G, Reingold J, Durrani S, Lewis GD, Newton-Cheh C, Scherrer-Crosbie M, Kaplan LM, Wang TJ. Effect of weight loss after weight loss surgery on plasma N-terminal pro-B-type natriuretic peptide levels. Am J Cardiol. 2010 Nov 15;106(10):1450-5. doi: 10.1016/j.amjcard.2010.06.076. PMID 21059435
- [Background] Bertoni AG, Wagenknecht LE, Kitzman DW, Marcovina SM, Rushing JT, Espeland MA; Brain Natriuretic Peptide Subgroup of the Look AHEAD Research Group. Impact of the look AHEAD intervention on NT-pro brain natriuretic peptide in overweight and obese adults with diabetes. Obesity (Silver Spring). 2012 Jul;20(7):1511-8. doi: 10.1038/oby.2011.296. Epub 2011 Sep 29. PMID 21959345
- [Background] Tsukamoto O, Fujita M, Kato M, Yamazaki S, Asano Y, Ogai A, Okazaki H, Asai M, Nagamachi Y, Maeda N, Shintani Y, Minamino T, Asakura M, Kishimoto I, Funahashi T, Tomoike H, Kitakaze M. Natriuretic peptides enhance the production of adiponectin in human adipocytes and in patients with chronic heart failure. J Am Coll Cardiol. 2009 Jun 2;53(22):2070-7. doi: 10.1016/j.jacc.2009.02.038. PMID 19477358
- [Background] Pivovarova O, Gogebakan O, Kloting N, Sparwasser A, Weickert MO, Haddad I, Nikiforova VJ, Bergmann A, Kruse M, Seltmann AC, Bluher M, Pfeiffer AF, Rudovich N. Insulin up-regulates natriuretic peptide clearance receptor expression in the subcutaneous fat depot in obese subjects: a missing link between CVD risk and obesity? J Clin Endocrinol Metab. 2012 May;97(5):E731-9. doi: 10.1210/jc.2011-2839. Epub 2012 Mar 14. PMID 22419733
- [Background] Miyashita K, Itoh H, Tsujimoto H, Tamura N, Fukunaga Y, Sone M, Yamahara K, Taura D, Inuzuka M, Sonoyama T, Nakao K. Natriuretic peptides/cGMP/cGMP-dependent protein kinase cascades promote muscle mitochondrial biogenesis and prevent obesity. Diabetes. 2009 Dec;58(12):2880-92. doi: 10.2337/db09-0393. Epub 2009 Aug 18. PMID 19690065
- [Background] Heinisch BB, Vila G, Resl M, Riedl M, Dieplinger B, Mueller T, Luger A, Pacini G, Clodi M. B-type natriuretic peptide (BNP) affects the initial response to intravenous glucose: a randomised placebo-controlled cross-over study in healthy men. Diabetologia. 2012 May;55(5):1400-5. doi: 10.1007/s00125-011-2392-1. Epub 2011 Dec 13. PMID 22159910
- [Background] Bordicchia M, Liu D, Amri EZ, Ailhaud G, Dessi-Fulgheri P, Zhang C, Takahashi N, Sarzani R, Collins S. Cardiac natriuretic peptides act via p38 MAPK to induce the brown fat thermogenic program in mouse and human adipocytes. J Clin Invest. 2012 Mar;122(3):1022-36. doi: 10.1172/JCI59701. Epub 2012 Feb 6. PMID 22307324
- [Background] Plante E, Menaouar A, Danalache BA, Broderick TL, Jankowski M, Gutkowska J. Treatment with brain natriuretic peptide prevents the development of cardiac dysfunction in obese diabetic db/db mice. Diabetologia. 2014 Jun;57(6):1257-67. doi: 10.1007/s00125-014-3201-4. Epub 2014 Mar 5. PMID 24595856
- [Background] Shankar SS, Shankar RR, Railkar RA, Beals CR, Steinberg HO, Kelley DE. Early Clinical Detection of Pharmacologic Response in Insulin Action in a Nondiabetic Insulin-Resistant Population. Curr Ther Res Clin Exp. 2015 Aug 14;77:83-9. doi: 10.1016/j.curtheres.2015.08.001. eCollection 2015 Dec. PMID 26543510
- [Background] Holmes SJ, Espiner EA, Richards AM, Yandle TG, Frampton C. Renal, endocrine, and hemodynamic effects of human brain natriuretic peptide in normal man. J Clin Endocrinol Metab. 1993 Jan;76(1):91-6. doi: 10.1210/jcem.76.1.8380606.
- [Background] Vila G, Grimm G, Resl M, Heinisch B, Einwallner E, Esterbauer H, Dieplinger B, Mueller T, Luger A, Clodi M. B-type natriuretic peptide modulates ghrelin, hunger, and satiety in healthy men. Diabetes. 2012 Oct;61(10):2592-6. doi: 10.2337/db11-1466. Epub 2012 Jun 14. PMID 22698919
- [Background] Mojiminiyi OA, Abdella NA, Al Arouj M, Ben Nakhi A. Adiponectin, insulin resistance and clinical expression of the metabolic syndrome in patients with Type 2 diabetes. Int J Obes (Lond). 2007 Feb;31(2):213-20. doi: 10.1038/sj.ijo.0803355. Epub 2006 Jun 6. PMID 16755284
- [Background] Timar R, Timar B, Degeratu D, Serafinceanu C, Oancea C. Metabolic syndrome, adiponectin and proinflammatory status in patients with type 1 diabetes mellitus. J Int Med Res. 2014 Oct;42(5):1131-8. doi: 10.1177/0300060514541829. Epub 2014 Jul 22. PMID 25053801